CLINICAL TRIAL: NCT07218679
Title: Clinical Trial on the Use of Stratafix Symmetric vs. Resorbable Monofilament for Closure of Large Median Laparotomy in Oncological Patients
Acronym: ONCOSTRAT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FIS-STRA-2024-01
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-07

CONDITIONS: Incisional Hernia After Midline Laparotomy
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Stratafix (Experimental): Midline laparotomy closure with Stratafix suture.
  Interventions: Device: Stratafix Suture
- PDS plus (Active Comparator): Midline laparotomy closure with PDS plus suture
  Interventions: Device: PDS plus suture

INTERVENTIONS:
Device: Stratafix Suture — Midline laparotomy closure using Stratafix vs PDS plus.
  Arms: Stratafix
Device: PDS plus suture — Midline laparotomy closure using PDS plus.
  Arms: PDS plus

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of using Stratafix (a type of symmetric, barbed, and coated suture) for abdominal wall closure in oncologic patients undergoing elective midline laparotomy, compared to the use of a monofilament suture following the Small Stitch technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age who will undergo midline laparotomy for oncologic resection of a retroperitoneal tumor or cytoreductive surgery for carcinomatosis of any origin.

Exclusion Criteria:

* Diagnosed incisional hernia.
* When the planned midline laparotomy is expected to be less than 20 cm.
* Patients with a BMI > 45 kg/m².
* Patients with abdominal aortic aneurysm.
* Patients with coagulopathy: previously diagnosed with von Willebrand disease, hemophilia, or idiopathic thrombocytopenic purpura.
* Patients with collagen disorders: previously diagnosed with Marfan syndrome, Ehlers-Danlos syndrome, homocystinuria, or scleroderma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Incisional hernia | 12 months
  Incisional hernia rate after midline laparotomy closure.

SECONDARY OUTCOMES:
Wound infection | 12 months.
  Compare the wound infection rate after midline laparotomy closure with Stratafix vs PDS plus.
Wound seroma | 12 months
  Compare the wound seroma rate after midline laparotomy closure with Stratafix vs PDS plus.
Hematoma | 12 months
  Compare the hematoma rate after midline laparotomy closure with Stratafix vs PDS plus.
Evisceration | 1 month
  Compare the evisceration rate after midline laparotomy closure with Stratafix vs PDS plus.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen del Rocio, Seville, Spain